CLINICAL TRIAL: NCT06569108
Title: A Randomized, Open-label Study to Evaluate the Efficacy and Safety of KN057 Injection Prophylaxis in Patients With Hemophilia A or B Without Inhibitors
Brief Title: Efficacy and Safety of KN057 Prophylaxis in Patients With Haemophilia A or B Without Inhibitors
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN057-A-302
Record Dates: First submitted 2023-12-30; First posted 2024-08-23 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A Without Inhibitor; Hemophilia B Without Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A：Experimental group (Experimental): Successfully screened participants in Part A will be randomly assigned to Experimental group versus Control group at a ratio of 2:1. Participants in Experimental group will receive KN057 prophylaxis through the main trial (26 weeks) and extension period (26 weeks) for total of approximately 1 year.
  Interventions: Drug: KN057
- Part A：Control group (Experimental): Successfully screened participants in Part A will be randomly assigned to Experimental group versus Control group at a ratio of 2:1. Participants in Control group will continue on-demand treatment with coagulation factor through the main trial for 26 weeks, in the extension period they will switch to prophylaxis treatment and receive KN057 for 26 weeks.
  Interventions: Drug: KN057
- Part B：Prophylaxis group (Experimental): Successfully screened participants in Part B will be nonrandomly assigned to Prophylaxis group. Participants in Prophylaxis group will continue prophylaxis with coagulation factor for the first 26 weeks (the factor period), then they will switch to prophylaxis with KN057 for the last 26 weeks (the KN057 period).
  Interventions: Drug: KN057

INTERVENTIONS:
Drug: KN057 — KN057 will be administered subcutaneously once a week.

SUMMARY:
The purpose of this study is to show that KN057 can prevent bleeds in patients with haemophilia A or B without inhibitors and is safe to use. Participants receiving on-demand treatment prior to screening will be randomly assigned to Experimental group or Control group at a ratio of 2:1 in Part A. Participants receiving prophylaxis prior to screening will be nonrandomly assigned to Prophylaxis group in Part B. Participants in Experimental group will receive KN057 prophylaxis for 52 weeks upon enrollment. Participants in Control group will first receive on-demand treatment for 26 weeks, then switch to KN057 prophylaxis for 26 weeks. Participants in Prophylaxis group will first receive prophylaxis with coagulation factor for 26 weeks, then switch to KN057 prophylaxis for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 12 to 70 years old at the time of signing informed consent (including the cut-off value), body weight ≥30 kg and BMI <28 kg/m^2 at screening;
2. Severe and moderately severe hemophilia A or hemophilia B (FVIII or FIX activity level ≤2%);
3. FVIII or FIX inhibitor test is negative (<0.6 BU/ml) or lower than the lower limit of laboratory normal values during the screening period;
4. There is no history of FVIII or FIX inhibitors in the past; or there has been an inhibitor, but it has been at least 5 years since successful immune tolerance induction therapy (ITI), and the inhibitor has not reappeared (a positive inhibitor was detected after successful ITI);
5. Use coagulation factor replacement therapy for no less than 100 exposure days before screening;
6. Have not used Anti-TFPI drugs before;
7. Be able and agree to elute the original hemophilia drugs.

Participants who are enrolled into Part A must also meet the following criteria:

1. ≥6 treated bleeding episodes within 26 weeks before screening;
2. Receiving on-demand treatment, non-standard prophylaxis, or standard prophylaxis no more than 12 weeks before screening;

Participants who are enrolled into Part B must also meet the following criteria:

Being on standard prophylaxis and maintaining it for more than 12 weeks (standard prophylaxis is defined as at least 80% compliance with a predetermined prophylaxis regimen).

Exclusion Criteria:

1. Have serious or poorly controlled chronic diseases or obvious systemic diseases;
2. Have a history of thromboembolic disease, or currently have symptoms or signs related to thromboembolic disease or being treated with thrombolytic/antithrombotic therapy;
3. Have high-risk factors for thrombosis: such as a history of coronary atherosclerotic disease, ischemic disease of important organs, vascular occlusive disease, autoimmune diseases with a high risk of thrombosis, or indwelling central venous catheter;
4. The presence of other inherited or acquired bleeding disorders other than hemophilia A and hemophilia B;
5. Known or suspected hypersensitivity to any constituent of the trial product or related products;
6. Have undergone major surgery (as determined by the investigator) within 3 months before screening, or have elective surgery planned during the study;
7. Used Emicizumab treatment within 6 months before screening;
8. Have received any gene therapy for hemophilia in the past;
9. Other factors that the investigator deems inappropriate for participating in this trial, such as the presence of concomitant diseases, treatment or examination abnormalities that affect the subject's safety during the trial or affect the interpretation of trial results.

Ages: 12 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Part A: Annualized bleeding rate (ABR) calculated based on treated spontaneous and traumatic bleeding episodes in Experimental group and Control group. | From Week 1 to Week 26, through the main trial.
  Treated bleeding refers to the use of coagulation factors for hemostatic treatment of the bleeding.
Part B: ABR calculated based on treated spontaneous and traumatic bleeding episodes in Prophylaxis group. | From Week 1 to Week 26, through the factor period. From Week 27 to Week 52, through the KN057 period.
  Treated bleeding refers to the use of coagulation factors for hemostatic treatment of the bleeding.

SECONDARY OUTCOMES:
ABR calculated based on bleeding episodes, treated spontaneous and traumatic bleeding episodes, treated spontaneous bleeding episodes, treated joint bleeding episodes, and treated target joint bleeding respectively in Experimental group. | From Week 1 to Week 52, through the main trial and extension period.
  Bleeding episodes includes spontaneous and/or traumatic bleeding episodes, excluding surgery/procedure-related bleeding episodes. Treated bleeding refers to the use of coagulation factors for hemostatic treatment of the bleeding. Target joint are those with spontaneous bleeding ≥3 times in the 6 months prior to screening.
ABR calculated based on bleeding episodes, treated spontaneous bleeding episodes, treated joint bleeding episodes, and treated target joint bleeding respectively in Experimental group, Control group and Prophylaxis group. | From Week 1 to Week 26. From Week 27 to Week 52.
  Bleeding episodes includes spontaneous and/or traumatic bleeding episodes, excluding surgery/procedure-related bleeding episodes. Treated bleeding refers to the use of coagulation factors for hemostatic treatment of the bleeding. Target joint are those with spontaneous bleeding ≥3 times in the 6 months prior to screening.
Proportion of participants with untreated bleeding episodes in Experimental group, Control group and Prophylaxis group. | From Week 1 to Week 26. From Week 27 to Week 52.
  Treated bleeding refers to the use of coagulation factors for hemostatic treatment of the bleeding.
The annual usage of on-demand treatment drugs (adjusted by body weight) in Experimental group and Control group. | From Week 1 to Week 26. From Week 27 to Week 52.
Change from baseline in Hemophilia Joint Health Score (HJHS) scores in Experimental group, Control group and Prophylaxis group. | From Week 1 to Week 26.
  Hemophilia Joint Health Scores (HJHS) is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 and 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Change in HJHS scores from baseline in Experimental group, from the 26th week in Control group, from baseline and the 26th week in Prophylaxis group. | From Week 1 to Week 52.
  Hemophilia Joint Health Scores (HJHS) is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 and 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Change from baseline in EuroQol 5 Dimensions 5 Level (EQ-5D-5L) in Experimental group, Control group and Prophylaxis group. | From Week 1 to Week 26.
  The EQ-5D-5L questionnaire is made up for 2 components, health state description and evaluation. In description part, health status is measured in terms of 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; every dimension contains 5 levels (5L): no difficulty, a little difficulty, moderate difficulty, severe difficulty, very severe difficulty/inability to perform. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Change in EQ-5D-5L from baseline in Experimental group, from the 26th week in Control group, from baseline and the 26th week in Prophylaxis group. | From Week 1 to Week 52.
  The EQ-5D-5L questionnaire is made up for 2 components, health state description and evaluation. In description part, health status is measured in terms of 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; every dimension contains 5 levels (5L): no difficulty, a little difficulty, moderate difficulty, severe difficulty, very severe difficulty/inability to perform. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Incidence of TEAE, TEAE related to the experimental drug and SAE. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
  TEAE refers to 'treatment emergent adverse event'. SAE refers to 'serious adverse event'.
Incidence of thromboembolic events, TMA and DIC. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
  TMA refers to 'thrombotic microangiopathy'. DIC refers to 'disseminated intravascular coagulation'.
Incidence of hypersensitivity type reactions. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
Incidence of injection site reactions. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
Incidence of clinically significant laboratory value abnormalities. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
Number of participants with clinically significant changes from baseline in physical exam. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
Number of participants with clinically significant changes from baseline in electrocardiograms. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
Number of participants with clinically significant changes from baseline in vital signs. | From the signing of informed consent to 4 weeks after the last dose of KN057 (the end of the trial), approximately 59 weeks in total.
KN057 plasma concentration. | From start of KN057 treatment (Week 1 for Experimental group, Week 26 for Control group and Prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for Experimental group and 30 weeks for Control group and Prophylaxis group.
  pharmacokinetics
Levels of Total TFPI. | From start of KN057 treatment (Week 1 for Experimental group, Week 26 for Control group and Prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for Experimental group and 30 weeks for Control group and Prophylaxis group.
  pharmacodynamics
Levels of Free TFPI. | From start of KN057 treatment (Week 1 for Experimental group, Week 26 for Control group and Prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for Experimental group and 30 weeks for Control group and Prophylaxis group.
  pharmacodynamics
Levels of prothrombin fragment 1+2 (PF1+2). | From start of KN057 treatment (Week 1 for Experimental group, Week 26 for Control group and Prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for Experimental group and 30 weeks for Control group and Prophylaxis group.
  pharmacodynamics
Incidence of anti-KN057 antibody (ADA) and neutralizing antibody (Nab). | From start of KN057 treatment (Week 1 for Experimental group, Week 26 for Control group and Prophylaxis group) to 4 weeks after the last dose of KN057, approximately 56 weeks for Experimental group and 30 weeks for Control group and Prophylaxis group.
  immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Doctor, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Jing Sun, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University; Hu Zhou, Doctor, Principal Investigator — Henan Cancer Hospital; Changcheng Zheng, Doctor, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital); Xielan Zhao, Doctor, Principal Investigator — Xiangya Hospital of Central South University; Lili Chen, Doctor, Principal Investigator — Tai Zhou First People's Hospital; Chenghao Jin, Doctor, Principal Investigator — Jiangxi Provincial People's Hopital; Yanping Song, Doctor, Principal Investigator — Xi'an Central Hospital; Yaming Xi, Doctor, Principal Investigator — LanZhou University; Zeping Zhou, Doctor, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University; Runhui Wu, Doctor, Principal Investigator — Beijing Children's Hospital; Jingyu Yan, Doctor, Principal Investigator — North China University of Science and Technology; Sujun Gao, Doctor, Principal Investigator — Bethune First Hospital of Jilin University; Wei Yang, Doctor, Principal Investigator — Shengjing Hospital of China University; Rong Zhou, Doctor, Principal Investigator — The Third People's Hospital of Chengdu; Ziqiang Yu, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University; Yun Chen, Doctor, Principal Investigator — Qianfoshan Hospital; Pingchong Lei, Doctor, Principal Investigator — Henan Provincial People's Hospital; Yinsuo Zheng, Doctor, Principal Investigator — Bao Ji Central Hospital; Peng Cheng, Doctor, Principal Investigator — First Affiliated Hospital of Guangxi Medical University; Jianwen Xiao, Doctor, Principal Investigator — Children's Hospital of Chongqing Medical University; Ruibin Huang, Doctor, Principal Investigator — The First Affiliated Hospital of Nanchang University; Hailiang Li, Doctor, Principal Investigator — The first affiliated hospital of jiangxi medical college; Shu Chen, Doctor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Xiong Zhang, Doctor, Principal Investigator — Maoming City People's Hospital; Jingyu Zhang, Doctor, Principal Investigator — The Second Hospital of Hebei Medical Hospital; Baolai Hua, Doctor, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University; Yanming Zhang, Doctor, Principal Investigator — Huai'an Second People'Hospital
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No